CLINICAL TRIAL: NCT05833672
Title: Single Arm Study of Neoadjuvant Immunotherapy Combined With Chemotherapy in Locally Advanced Colon Cancers
Brief Title: Neoadjuvant Immunotherapy in Locally Advanced Colon Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: fan li (Other)
Responsible Party: Sponsor-Investigator, fan li, Prof., Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NICO-D
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Colon Cancer; Immunotherapy
Keywords: Immunotherapy; Colon Cancer; neoadjuvant; Terelizumab; Multi-omics analysis
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Locally Advanced Colon Cancers (Experimental): Cycle 1 to Cycle 2 CapeOX + Terelizumab therapy(Day 1 through Day 21)
  Interventions: Drug: Terelizumab; Drug: CapeOx

INTERVENTIONS:
Drug: Terelizumab — q3w Terelizumab 200mg on day 1 of each cycle
Drug: CapeOx — Oxaliplatin(130mg/m2) on day 1 of each cycle and Capecitabine:Dose of 1000mg/m2,14days

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of neoadjuvant immunotherapy combined with chemotherapy before colonic resection in patients with locally advanced colon cancers

DETAILED DESCRIPTION:
The trial is designed as an investigator-initiated, single center, prospective, single arm phase II study in patients with locally advanced colon cancers scheduled for intended curative surgery to determine the efficacy of immunotherapy using tislelizumab in the neoadjuvant setting. Patients will receive CapeOX + Terelizumab therapy(Day 1 through Day 21) following diagnosis. After 3 weeks a re-evaluation (to assess tumor response) will be performed, followed by standard surgery for resection of the tumor. Surgery will therefore be performed within 3 to 5 weeks after 2 cycle of neoadjuvant combined immunotherapy.. The patients will be followed as per the standard Danish guidelines with CT scans at 1 and 3 years after surgery. The specimen collected by surgery and clinical data will be collected . We use Integrative omics analysis to establish a clinical efficacy prediction model by means of bioinformatics to prospectively judge the efficacy and guide the follow-up individualized and accurate treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patients are able to understand and voluntarily sign the written informed consent, which must be signed prior to the implementation of the designated research procedures required by the study.
2. The age at the time of signing the informed consent form (ICF) is ≥ 18 years old, both male and female.
3. Locally advanced colonic adenocarcinoma (clinical stage T3-4N0M0 or T1-4N+M0 ) were diagnosed by comprehensive evaluation.
4. The patients are willing to provide fresh tissue for biomarker analysis, and the tissue samples provided are of sufficient quality to evaluate the status of biomarkers. If sufficient tissue is not provided, repeated sampling may be required.
5. The patient has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
6. The expected survival time was ≥ 3 months.
7. The patient has adequate organs function. 1)The patient has adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥1.5*10^9/L, hemoglobin ≥90g/L (5.58 mmol/L), and platelets ≥100*10^9/L.

2)The patient has adequate renal function as defined by a serum creatinine ≤1.5 times the ULN, or creatinine clearance (measured via 24-hour urine collection) ≥50 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed).

3)The patient has adequate hepatic function as defined by a total bilirubin ≤1.5 mg/dL (25.65 μmol/L), and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times the upper limit of normal (ULN; or 5.0 times the ULN in the setting of liver metastases).

4)The patient must have adequate coagulation function as defined by international normalized ratio (INR) ≤1.5 8.Within 7 days before the first administration, women of childbearing age must confirm that the serum pregnancy test is negative and agree to use effective contraceptives during the study period and within 180 days after the last administration. In this program, women of childbearing age are defined as sexually mature women:

1. No hysterectomy or bilateral ovariectomy
2. Natural menopause does not last for 24 months (amenorrhea after cancer treatment does not rule out fertility) (that is, menstruation occurs at any time in the previous 24 months).

9.For male patients whose sexual partners are women of childbearing age, they must agree to use effective contraception during the study drug use and within 180 days after the last administration.

Exclusion Criteria:

1. Palliative local treatment was given to non-target lesions within 2 weeks before the first administration, and systemic non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, etc.) was received within 2 weeks before the first administration. Chinese herbal medicine or proprietary Chinese medicine with anti-tumor indications was received within 2 weeks before the first administration.
2. The patient has previously received immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as antibodies against ICOS, CD40, CD137, GITR, OX40 targets, etc.), immune cell therapy, etc. any treatment aimed at the immune mechanism of tumor.
3. There was a history of gastrointestinal perforation and gastrointestinal fistula within 6 months before the first administration. If the perforation or fistula has been removed or repaired, and the disease has been judged by the researchers to recover or remission, it may be allowed to join the group.
4. Active or previously recorded inflammatory bowel disease (such as Crohn's disease or ulcerative colitis). Unable to swallow, malabsorption syndrome, or uncontrollable nausea, vomiting, diarrhea or other gastrointestinal diseases that seriously affect drug use and absorption.
5. There were active malignant tumors in the past 3 years, except for tumors that participated in the study and local tumors that had been cured. such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, breast cancer in situ, localized prostate cancer and so on.
6. A history of allergy to study drug components or a history of severe hypersensitivity reaction to any monoclonal antibody.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 6 months
  Pathological complete response will be evaluated with American Joint Committee on Cancer (AJCC) Cancer Staging
ORR (objective response rate) | 6 months
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor

SECONDARY OUTCOMES:
Major pathologic response (MPR) | 6 months
  It is defined as residual tumors less than 10% after neoadjuvant immunotherapy and(or) chemotherapy
Overall survival (OS) | 2 years
  Time from study entry to death from any cause.
Disease-free survival (DFS) | 2 years
  Time from study entry to disease recurrence or patient death due to disease progression
R0 resection rate | 6 months
  Rate of microscopically margin-negative resection

CONTACTS AND LOCATIONS:
Locations (1):
- Daping hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided